CLINICAL TRIAL: NCT05107817
Title: Catching and Throwing Exercises to Improve Reactive Balance: A Randomized Controlled Trial Protocol for the Comparison of Aquatic and Dry-land Training Environments
Brief Title: Aquatic Exercise and Reactive Balance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eadric Bressel (Other)
Responsible Party: Sponsor-Investigator, Eadric Bressel, Professor, Utah State University
Organization: Utah State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12227
Record Dates: First submitted 2021-10-14; First posted 2021-11-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Aging; Aged; Accidental Falls; Postural Balance; Exercise; Exercise Therapy
Keywords: Reactive balance; Aquatic exercise; Aquatic therapy; Fall prevention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aquatic Exercise group (Experimental): Participants will engage in a single session of training consisting of 120 repetitions of a ball throwing and catching task in water.
  Interventions: Other: Exercise intervention
- Land Exercise group (Active Comparator): Participants will engage in a single session of training consisting of 120 repetitions of a ball throwing and catching task on dry land.
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Other: Exercise intervention — A ball catching and throwing exercise.

SUMMARY:
The present clinical trial aims to identify if skills acquired during aquatic exercise are more effectively transferred to a reactive balance task than land exercise. This study is designed as a double-blinded, randomized controlled clinical trial. Forty-four older adults aged 60 years or above who meet the eligibility criteria will be recruited and randomized into an aquatic exercise group or land exercise group. Each group will participate in the same balance training exercise during a single session that includes a ball throwing and catching task. A modified lean-and-release test will be implemented on land immediately before, after, and one week after the training session. The outcomes will include reaction time, rapid response accuracy, and mini-BESTest scores obtained from stepping and grasping reactions.

DETAILED DESCRIPTION:
During the modified lean-and-release test, there are two possible settings: 1) the leg block is placed in front of both legs, and a safety handle is uncovered; or 2) the leg block is removed, and the safety handle is covered. The leg block and handle cover will be controlled via computer-triggered, servo motors. The testing session will be comprised of three blocks: 1) REACH (grasping a safety handle using their right hand while maintaining both feet fixed), 2) STEP (stepping forward using any leg), and 3) RANDOM (random variations of STEP and REACH).

ELIGIBILITY:
Inclusion Criteria:

* Ability to stand using a double-leg stance for one minute of time
* Ability to walk independently
* Normal or corrected to normal vision
* Normal or corrected to normal hearing based on a qualitative assessment

Exclusion Criteria:

* Any neurological or musculoskeletal disorders that may inhibit the participation in the training and testing protocols
* A concussion within the past one year before the participation
* Any cognitive deficiencies (e.g., memory, concentration, or attention disorder)
* One or more 'yes' answered on the Physical Activity Readiness Questionnaire (PAR-Q)
* Fear of water

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Reaction time measures (REACH) | Immediately before the intervention. Duration of each assessment will be 15 minutes.
  Hand contact time during REACH following the cable release will be calculated.
Reaction time measures (STEP1) | Immediately before the intervention. Duration of each assessment will be 15 minutes.
  Foot-off time during STEP following the cable release will be calculated.
Reaction time measures (STEP2) | Immediately before the intervention. Duration of each assessment will be 15 minutes.
  Foot contact time during STEP following the cable release will be calculated.
Rapid response accuracy | Immediately before the intervention. Duration of each assessment will be 15 minutes.
  For the RANDOM block, response accuracy, defined as the percentage of accurate responses, will be calculated. To represent a composite measure of accuracy and speed of response, rapid response accuracy will be calculated using the ratio of response accuracy to the reaction time (%/ms). Foot-off and hand contact data will be used for the calculation.
Mini-Balance Evaluation Systems Test | Immediately before the intervention. Duration of each assessment will be 15 minutes.
  During the REACH, STEP, and RANDOM blocks, the quality of the compensatory reactions will be scored using the Reactive Postural Control section of the Mini-Balance Evaluation Systems Test. The scores will be ranged from 0 (worst) to 2 (best).
Reaction time measures (REACH) | Immediately after the intervention. Duration of each assessment will be 15 minutes.
  Hand contact time during REACH following the cable release will be calculated.
Reaction time measures (STEP1) | Immediately after the intervention. Duration of each assessment will be 15 minutes.
  Foot-off time during STEP following the cable release will be calculated.
Reaction time measures (STEP2) | Immediately after the intervention. Duration of each assessment will be 15 minutes.
  Foot contact time during STEP following the cable release will be calculated.
Rapid response accuracy | Immediately after the intervention. Duration of each assessment will be 15 minutes.
  For the RANDOM block, response accuracy, defined as the percentage of accurate responses, will be calculated. To represent a composite measure of accuracy and speed of response, rapid response accuracy will be calculated using the ratio of response accuracy to the reaction time (%/ms). Foot-off and hand contact data will be used for the calculation.
Mini-Balance Evaluation Systems Test | Immediately after the intervention. Duration of each assessment will be 15 minutes.
  During the REACH, STEP, and RANDOM blocks, the quality of the compensatory reactions will be scored using the Reactive Postural Control section of the Mini-Balance Evaluation Systems Test. The scores will be ranged from 0 (worst) to 2 (best).
Reaction time measures (REACH) | One week after the intervention. Duration of each assessment will be 15 minutes.
  Hand contact time during REACH following the cable release will be calculated.
Reaction time measures (STEP1) | One week after the intervention. Duration of each assessment will be 15 minutes.
  Foot-off time during STEP following the cable release will be calculated.
Reaction time measures (STEP2) | One week after the intervention. Duration of each assessment will be 15 minutes.
  Foot contact time during STEP following the cable release will be calculated.
Rapid response accuracy | One week after the intervention. Duration of each assessment will be 15 minutes.
  For the RANDOM block, response accuracy, defined as the percentage of accurate responses, will be calculated. To represent a composite measure of accuracy and speed of response, rapid response accuracy will be calculated using the ratio of response accuracy to the reaction time (%/ms). Foot-off and hand contact data will be used for the calculation.
Mini-Balance Evaluation Systems Test | One week after the intervention. Duration of each assessment will be 15 minutes.
  During the REACH, STEP, and RANDOM blocks, the quality of the compensatory reactions will be scored using the Reactive Postural Control section of the Mini-Balance Evaluation Systems Test. The scores will be ranged from 0 (worst) to 2 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Eadric Bressel, Principal Investigator — Utah State University

IPD SHARING:
Plan to Share IPD: No
Any individual participant data collected in this study will not be shared with other researchers to follow the HIPAA Privacy Rule.

REFERENCES:
- [Background] Bolton DAE, Mansour M. A Modified Lean and Release Technique to Emphasize Response Inhibition and Action Selection in Reactive Balance. J Vis Exp. 2020 Mar 19;(157):10.3791/60688. doi: 10.3791/60688. PMID 32250359
- See also: Related Info — https://www.jove.com/t/60688/a-modified-lean-release-technique-to-emphasize-response-inhibition